CLINICAL TRIAL: NCT01361945
Title: A Phase I/ II, Multi-center, Open-label Study, to Evaluate the Efficacy of AUY922 in Combination With Lapatinib With Letrozole in Postmenopausal Patients With Locally Advanced or Metastatic ER+ , HER2 + Breast Cancer
Brief Title: AUY922 With Lapatinib and Letrozole for ER+ HER2+ Advanced Breast Cancer
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed due to no enrollment
Sponsor: Texas Tech University Health Sciences Center, El Paso (Other)
Responsible Party: Principal Investigator, Zeina Nahleh, Professor, Texas Tech University Health Sciences Center, El Paso
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAUY922ZN11
Record Dates: First submitted 2011-05-24; First posted 2011-05-27 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2015-12

CONDITIONS: Breast Cancer; Metastatic Breast Cancer; HER-2 Positive Breast Cancer; ER Positive Breast Cancer
Keywords: ER+; HER2+; Breast
MeSH Terms: conditions — Breast Neoplasms | interventions — 5-(2,4-dihydroxy-5-isopropylphenyl)-4-(4-morpholin-4-ylmethylphenyl)isoxazole-3-carboxylic acid ethylamide; Infusion Pumps

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AUY922 (Experimental): Single Arm
  Interventions: Drug: AUY922

INTERVENTIONS:
Drug: AUY922 — AUY 922 is given intravenously weekly; letrozole and lapatinib are given orally
  Other Names: Intravenous drug

SUMMARY:
The purpose of this study is to find out what effects, administering infusions of AUY922 with hormonal therapy (letrozole) and oral targeted drug (lapatinib) will have on the patients with advanced breast cancer known as ER+ HER2 +.

DETAILED DESCRIPTION:
The dose and schedule of AUY922 is the MTD dose identified in the phase I, given as 1 hour infusion weekly.

The Phase II component will have a 2 stage design single arm design. (Section 9.0). Overall response rate (ORR) is the primary endpoint. Estimated N=40 (12 in first stage) .A total of 39 response-evaluable participants is required. In the first stage, 12 response-evaluable participants will be accrued; if there are 3 or fewer CR+PRs, the study will stop for futility. There is a 55% probability of stopping early if, in fact, the ORR is 28%. If there are 4 or more CR+PRs, the study will proceed to the second stage and an additional 27 response-evaluable participants will be accrued. We will accrue 1 additional patient (then the needed 39 to account for attrition)

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years
* Able to sign Informed Consent
* Patients must have the following laboratory values:

Absolute Neutrophil Count (ANC) 1.5x109/L Hemoglobin (Hgb) 9 g/dl Platelets (plt) 100x109/L

* Potassium within normal limits
* Total calcium (corrected for serum albumin) and Phosphorus within normal limits
* Magnesium above LLN or correctable with supplements
* AST/SGOT and ALT/SGPT ≤ 1.5 x Upper Limit of Normal (ULN) if AP > 2.5 ULN
* AST/SGOT and ALT/SGPT ≤ 2.5 x Upper Limit of Normal (ULN) if AP ≤ 5.0 x ULN if
* Serum bilirubin 1.5 x ULN
* Serum creatinin 1.5 x ULN or 24-hour clearance 50 ml/min
* Negative serum pregnancy test. The serum pregnancy test must be obtained prior to the first administration of AUY922 (≤ 72 hours prior to dosing) in all pre-menopausal women and women <2 years after the onset of menopause
* Histologically confirmed HER2 + and ER+ or PR + (i.e., HR+) Postmenopausal women with Metastatic breast cancer or resistant locally advanced breast cancer.
* Stage of disease (stage IIIb/c not responding or progressing to standard therapy with trastuzumab) or stage IV receiving first line treatment in the metastatic setting . All patients should have documented clinical progression prior to entering study
* Prior chemotherapy for metastatic stage IV disease is prohibited for patients enrolled in phase II, but allowed up to 3 lines for patients enrolled in Phase I. Prior neoadjuvant/adjuvant chemotherapy, antiestrogens, and radiotherapy are allowed. Adjuvant hormonal therapy including aromatase inhibitors are permitted in the adjuvant, neoadjuvant or metastatic setting if discontinued at least two weeks prior to starting study treatment. Trastuzumab is permitted in the adjuvant, neoadjuvant or metastatic setting if discontinued at least 4 weeks prior to study treatment
* Patients must have at least one measurable lesion as defined by RECIST. Irradiated lesions and non-measurable disease are only evaluable for disease progression
* Patients must have tumors that carry HER-2 gene amplifications as determined by (i) fluorescence in situ hybridization (FISH) or (ii) overexpression of HER-2 protein 3+ level assessed by immunohistochemistry. Patients who have previously been treated with trastuzumab must be off treatment at least 6 weeks prior to starting study treatment.
* World Health Organization (WHO) Performance Status of < 1
* Life expectancy of > 12 weeks

Exclusion Criteria:

* Unresolved diarrhea ≥ CTCAE (v4.02) grade 1
* Pregnant or lactating women
* Impaired cardiac function, including any one of the following:
* History (or family history) of long QT syndrome
* Mean QTc ≥ 450 msec on baseline ECG
* History of clinically manifested ischemic heart disease ≤ 6 months prior to study start or History of heart failure or left ventricular (LV) dysfunction (LVEF ≤ 45%) by MUGA or ECHO or arrythmia
* Patients known to be HIV positive. Testing is not required in the absence of clinical signs and symptoms suggesting HIV infection.
* Known hypersensitivity to any of the study drugs or their excipients
* Participation in another clinical study within 30 days before first study treatment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | 2 years
  noted by tumor response using RECIST criteria

CONTACTS AND LOCATIONS:
Overall Officials: Zeina Nahleh, M.D., Principal Investigator — Texas Tech University Health Sciences Center, El Paso

IPD SHARING:
Plan to Share IPD: No
the study has not been completed